CLINICAL TRIAL: NCT03417934
Title: Effects of Hip Distraction Without a Perineal Post on Venous Blood Flow and Peripheral Nerve Conduction During Hip Arthroscopic Procedures Clinical Protocol: Prospective Study
Brief Title: Effects of Hip Distraction Without a Perineal Post on Venous Blood Flow and Peripheral Nerve Conduction
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0930
Record Dates: First submitted 2018-01-19; First posted 2018-01-31 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Hip Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hip Arthroscopy Procedure — The purpose of this pilot study is to evaluate the effects of hip distraction without a perineal post on the lower extremity during hip arthroscopic procedures by peri-operative monitoring of various prognostic markers for venous, nerve and tissue injury.

SUMMARY:
The purpose of this pilot study is to evaluate the effects of hip distraction without a perineal post on the lower extremity during hip arthroscopic procedures by peri-operative monitoring of various prognostic markers for venous, nerve and tissue injury.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the effects of hip distraction without a perineal post on the lower extremity during hip arthroscopic procedures by peri-operative monitoring of various prognostic markers for venous, nerve and tissue injury. The data from this exploratory study can be used to help develop estimates of the proportions of patients who experience significant venous/nerve/tissue compromise in the lower extremity as a result of the application of traction forces necessary to achieve hip joint distraction, and may serve as a basis for sample size planning in future studies comparing the effects of various methods of hip distraction techniques during hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusively
* Has elected to undergo a standard hip arthroscopic procedure that is expected to require access to the central compartment of the hip joint (bilateral hip enrollment is allowed)
* Is able to give voluntary, written informed consent to participate in this clinical investigation and has signed an informed consent document

Exclusion Criteria:

* Any major systemic or lower extremity trauma, or any preexisting medical condition/illness that represents a contraindication for hip arthroscopy surgery
* Significant peripheral vascular disease characterized by diminished dorsalis pedis or tibial pulse
* Significant peripheral neuropathy demonstrated by nerve conduction velocity test
* Preoperative use of statins or other medications known to elevate serum CPK-MM levels within one week of surgery
* Total hip replacement of the indicated hip(s)
* History of substance abuse within past 12 months (this includes any chronic narcotic use)
* Any significant psychological disturbance past or present, psychotic or neurotic, that could impair the informed consent process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population description is to include male or female subjects between the ages of 18 and 65 years, inclusively, with an election to undergo a standard hip arthroscopic procedure that is expected to require access to the central compartment of the hip joint (bilateral hip enrollment is allowed).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Intra-operative application of hip distraction without a perineal post to the lower extremity during hip arthroscopy procedures. | 12 Days
  Routine intra-operative application of hip distraction without a perineal post to the lower extremity during hip arthroscopy procedures will result in significant blood flow alterations as measured by Doppler ultrasonography.

SECONDARY OUTCOMES:
Pre- and post-operative screening for DVT. | 12 Days
  Pre- and post-operative screening for Deep Vein Thrombosis (DVT) using the D-Dimer assay test is correlative with intra-operative venous blood flow measurements.
Estimate the amount of tissue/muscle damage associated with hip arthroscopy procedures. | 12 Days
  To quantitatively estimate the amount of tissue/muscle damage associated with hip arthroscopy procedures using creatine phosphokinase (CPK-MM) serum levels as a prognostic marker.
Blood Flow Alterations | 12 Days
  To determine whether routine intra-operative application of hip distraction without a perineal post to the lower extremity during hip arthroscopy procedures results in significant blood flow alterations as measured by significant changes in peripheral nerve conduction as measured by Somatosensory Evoked Potentials (SSEP).

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei-Dan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Hip Preservation Center, Orthopedic Department, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrd JW, Chern KY. Traction versus distension for distraction of the joint during hip arthroscopy. Arthroscopy. 1997 Jun;13(3):346-9. doi: 10.1016/s0749-8063(97)90032-3. PMID 9195032
- [Background] Kelly BT, Buly RL. Hip arthroscopy update. HSS J. 2005 Sep;1(1):40-8. doi: 10.1007/s11420-005-0105-3. PMID 18751808
- [Background] Smart LR, Oetgen M, Noonan B, Medvecky M. Beginning hip arthroscopy: indications, positioning, portals, basic techniques, and complications. Arthroscopy. 2007 Dec;23(12):1348-53. doi: 10.1016/j.arthro.2007.06.020. Epub 2007 Oct 3. PMID 18063180
- [Background] Eriksson E, Arvidsson I, Arvidsson H. Diagnostic and operative arthroscopy of the hip. Orthopedics. 1986 Feb;9(2):169-76. doi: 10.3928/0147-7447-19860201-07. PMID 3960759
- [Background] Mei-Dan O, Kraeutler MJ, Garabekyan T, Goodrich JA, Young DA. Hip Distraction Without a Perineal Post: A Prospective Study of 1000 Hip Arthroscopy Cases. Am J Sports Med. 2018 Mar;46(3):632-641. doi: 10.1177/0363546517741704. Epub 2017 Dec 15. PMID 29244523
- [Background] Baber YF, Robinson AH, Villar RN. Is diagnostic arthroscopy of the hip worthwhile? A prospective review of 328 adults investigated for hip pain. J Bone Joint Surg Br. 1999 Jul;81(4):600-3. doi: 10.1302/0301-620x.81b4.8803. PMID 10463728
- [Background] Byrd JW. Chapter 16. Complications associated with hip arthroscopy. In Operative Hip Arthroscopy (2nd edition); Springer: New York, 2005.
- [Background] Ilizaliturri VM Jr. Complications of arthroscopic femoroacetabular impingement treatment: a review. Clin Orthop Relat Res. 2009 Mar;467(3):760-8. doi: 10.1007/s11999-008-0618-4. Epub 2008 Nov 19. PMID 19018604
- [Background] McCarthy JC, Lee JA. Hip arthroscopy: indications, outcomes, and complications. Instr Course Lect. 2006;55:301-8. PMID 16958465
- [Background] Bushnell BD, Anz AW, Bert JM. Venous thromboembolism in lower extremity arthroscopy. Arthroscopy. 2008 May;24(5):604-11. doi: 10.1016/j.arthro.2007.11.010. Epub 2008 Jan 7. PMID 18442695
- [Background] Bushnell BD, Dahners LE. Fatal pulmonary embolism in a polytraumatized patient following hip arthroscopy. Orthopedics. 2009 Jan;32(1):56. doi: 10.3928/01477447-20090101-01. PMID 19226026
- [Background] Jones SC, Fernau R, Woeltjen BL. Use of somatosensory evoked potentials to detect peripheral ischemia and potential injury resulting from positioning of the surgical patient: case reports and discussion. Spine J. 2004 May-Jun;4(3):360-2. doi: 10.1016/j.spinee.2003.08.023. PMID 15125862
- [Background] Chung I, Glow JA, Dimopoulos V, Walid MS, Smisson HF, Johnston KW, Robinson JS, Grigorian AA. Upper-limb somatosensory evoked potential monitoring in lumbosacral spine surgery: a prognostic marker for position-related ulnar nerve injury. Spine J. 2009 Apr;9(4):287-95. doi: 10.1016/j.spinee.2008.05.004. Epub 2008 Aug 5. PMID 18684675
- [Background] Pereles TR, Stuchin SA, Kastenbaum DM, Beric A, Lacagnino G, Kabir H. Surgical maneuvers placing the sciatic nerve at risk during total hip arthroplasty as assessed by somatosensory evoked potential monitoring. J Arthroplasty. 1996 Jun;11(4):438-44. doi: 10.1016/s0883-5403(96)80034-9. PMID 8792251
- [Background] Demers C, Marcoux S, Ginsberg JS, Laroche F, Cloutier R, Poulin J. Incidence of venographically proved deep vein thrombosis after knee arthroscopy. Arch Intern Med. 1998 Jan 12;158(1):47-50. doi: 10.1001/archinte.158.1.47. PMID 9437378
- [Background] Delis KT, Hunt N, Strachan RK, Nicolaides AN. Incidence, natural history and risk factors of deep vein thrombosis in elective knee arthroscopy. Thromb Haemost. 2001 Sep;86(3):817-21. PMID 11583313
- [Background] Wells PS, Anderson DR, Rodger M, Forgie M, Kearon C, Dreyer J, Kovacs G, Mitchell M, Lewandowski B, Kovacs MJ. Evaluation of D-dimer in the diagnosis of suspected deep-vein thrombosis. N Engl J Med. 2003 Sep 25;349(13):1227-35. doi: 10.1056/NEJMoa023153. PMID 14507948
- [Background] Ennis RS. Deep Venous Thrombosis Prophylaxis in Orthopedic Surgery. eMedicine; June 12, 2009. http)/emedicine.medscape.com/article/1268573-overview. Webpage accessed December 8, 2009.
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Merritt CR. Ultrasound safety: what are the issues? Radiology. 1989 Nov;173(2):304-6. doi: 10.1148/radiology.173.2.2678243. No abstract available.
- [Background] BlueCross BlueShield of Texas. Intra-operative Neurophysiologic Monitoring (Sensory-Evoked Potentials, Motor Evoked Potentials, EMG Monitoring). Medical Policy Bulletin (MED 205.011); Effective Date: 12/11/03.
- [Background] Martin HD, Palmer IJ, Champlin K, Kaiser B, Kelly B, Leunig M. Physiological changes as a result of hip arthroscopy performed with traction. Arthroscopy. 2012 Oct;28(10):1365-72. doi: 10.1016/j.arthro.2012.04.139. Epub 2012 Aug 21. PMID 22920287